CLINICAL TRIAL: NCT03990441
Title: Analgesic Efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) Versus Placebo During the First Stage of Labor. Double-blind Randomized Clinical Trial
Brief Title: Analgesic Efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) Versus Placebo During the First Stage of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: Hospital General Universitario de Castellón (Other)
Responsible Party: Principal Investigator, Manuel José Sos Gallen, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOS1
Record Dates: First submitted 2019-05-28; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Transcutaneous Electric Nerve Stimulation; Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): TENS application using the TensMed S82 (Enraf Nonius). Current parameters: balanced symmetric biphasic square waveform, continuous stimulation, frequency 80 Hz, pulse duration modulated between 250 and 290 μs, modulation time 5 seconds. Self-adhesive electrodes of 50 x 90 mm applied paravertebrally to 2 cm. of the spinous apophysis. Use of two channels with independent intensity (mA): electrodes of the first channel applied at level T10-L1 and second channel ones at level S2-S4. Maximum intensity without reaching pain, increasing the intensity throughout the application to maintain this level. Start of the intervention when the woman expresses pain. End of the intervention when neuraxial anesthesia is applied (if the woman demands it) or after delivery.
  Interventions: Device: TENS
- Placebo (Placebo Comparator): Same application as Intervention, but using 0,1 mA as fixed intensity on both channels.
  Interventions: Device: TENS Placebo

INTERVENTIONS:
Device: TENS — TENS application using the TensMed S82 (Enraf Nonius). Current parameters: balanced symmetric biphasic square waveform, continuous stimulation, frequency 80 Hz, pulse duration modulated between 250 and 290 μs, modulation time 5 seconds. Self-adhesive electrodes of 50 x 90 mm applied paravertebrally to 2 cm. of the spinous apophysis. Use of two channels with independent intensity (mA): electrodes of the first channel applied at level T10-L1 and second channel ones at level S2-S4. Maximum intensity without reaching pain, increasing the intensity throughout the application to maintain this level. Start of the intervention when the woman expresses pain. End of the intervention when neuraxial anesthesia is applied (if the woman demands it) or after delivery.
  Arms: Intervention
Device: TENS Placebo — Same application as Intervention, but using 0,1 mA as fixed intensity on both channels.
  Arms: Placebo

SUMMARY:
This study seeks to verify the analgesic efficacy of TENS during the first stage of labor applying TENS parameters that, according to with the evidence, can be effective for this application and discarding the placebo effect according to the methodological recommendations.

DETAILED DESCRIPTION:
TENS is a non-pharmacological alternative for pain control during labor. Although it's a method that has been used for decades, there is not enough evidence on its efficacy, so it's considered ineffective in the Spanish and British guidelines of clinical practice. The present study seeks to verify the analgesic efficacy of TENS by applying the electrodes in the spinal nerve roots associated with labor pain and using conventional TENS with parameters that, according to the evidence, may be effective for this application.

ELIGIBILITY:
Inclusion Criteria:

- Women attending routinary fetal monitoring before labor

Exclusion Criteria:

* Multiparous
* Scheduled cesarean
* Implantable Cardioverter Defibrillator (ICD) or pacemaker
* Epilepsy
* Fetal malformation
* Language barrier

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measure | Start of intervention, each 30 minutes during intervention, end of intervention (when neuraxial anesthesia is applied -if the woman demands it- or after delivery, assessed up to 10 hours from intervention's start).
  Self reported pain intensity. Score 0-10 (0 = no pain, 10 = pain as bad as can be), using a 0-10 pain scale combined with colored faces pain scale, for measuring the change of pain.

SECONDARY OUTCOMES:
TENS satisfaction | At leaving the labor room, assessed up to 3 hours after delivery.
  Self reported interest on use of TENS on future deliveries. Score 0-10 (0 = no way, 10 = absolutely necessary)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel José Sos Gallén, PT, PGCert, Study Director — Cardenal Herrera University
Locations (1):
- Hospital General Universitario de Castellón, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No